CLINICAL TRIAL: NCT06580678
Title: A Clinical Study to Evaluate Physiologic Dentin Regeneration When KH001 Was Administration to Erupted Wisdom Tooth With Dentin Caries
Brief Title: A Study to Evaluate Physiologic Dentin Regeneration and Safety of KH001 in the Administration of Erupted Wisdom Tooth With Dentin Caries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Byoung-Moo Seo (Other)
Collaborators: HysensBio Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, Byoung-Moo Seo, Principal Investigator, Seoul National University Dental Hospital
Organization: Seoul National University Dental Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KH-002-I201
Record Dates: First submitted 2024-08-11; First posted 2024-08-30 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Dentin Caries
Keywords: Wisdom Tooth; Dentin Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): KH001
  Interventions: Drug: KH001
- Group B (Placebo Comparator): Water for Injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KH001 — topical application of KH001
  Arms: Group A
Drug: Placebo — topical application of Water for Injection
  Arms: Group B

SUMMARY:
The purpose of this study is to evaluate physiologic dentin regeneration and safety of KH001 in the administration of erupted wisdom tooth with dentin caries

DETAILED DESCRIPTION:
The design is a single site, double-blind, randomized study. Phase 2 study to evaluate physiologic dentin regeneration and safety of KH001. The total duration of the study will be approximately 5 to 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Is between 19 and 35 of age by the time of the screening
* Has signed written informed consent in the study
* Subject who either have no pain in the affected tooth, or can endure pain until the day of tooth extraction

Exclusion Criteria:

* Is allergic to the active ingredient or other ingredients used in the investigational product
* Have participated in another clinical study within 30 days from screening visit and have a history of administration/application of investigational product/device
* Is judged by the investigator as ineligible for participation for other reasens

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of physiological dentin formation | Week 5
  Histological analysis after wisdom tooth extraction by histological analysis

SECONDARY OUTCOMES:
Adverse Events | Up to 9 weeks
  The adverse event name, onset date, resolution date, and other relevant details will be recorded until end of visit.
Oral soft/hard tissue examination | Up to 9 weeks
  Evaluation of oral condition by referring to maximum probing depth.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Dental Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No